CLINICAL TRIAL: NCT03297892
Title: Etat de santé Des Patients Suivis Pour Une Maladie de Cushing Dans la région Grand-Ouest de 1990 à 2015
Brief Title: Health Status of the Patients Followed for a Disease of Cushing in the Region Large-West of 1990 to 2015
Acronym: CUSHING
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CUSHING RB (15.217)
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Cushing Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cushing's disease is a rare disease that can reduce patients' expectations or quality of life, and for which predictive factors for cardiovascular mortality and recurrence are not well defined.

The primary objective is to determine the rates of remission and recurrence of patients with Cushing's disease diagnosed between 1990 and 2015 in the French region of the West (Angers, Brest, Nantes, Rennes, Poitiers , Tours) focusing on remission particularly at two periods : that after the first pituitary surgery and that on the day of the last news.

The secondary objective is to study the possible prediction of clinical and biological data perioperative of remission and recurrence during follow-up.

DETAILED DESCRIPTION:
Investigators are interested in the prevalence of complications of the pathology (cardiovascular, metabolic, neuropsychological, infectious, rheumatological, etc.) within this cohort, the mortality rate, the rate of remission and recurrence and the quality of life history using the history of patient illness and a questionnaire.

All patients over the age of 18 years at the time of inclusion, formerly or currently being monitored for Cushing's disease diagnosed between January 1, 1990 and December 31, 2015, in one of the six university centers in the West part of France can be included.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18 at inclusion,
* formerly or currently being followed for Cushing's disease diagnosed between 1 January 1990 and 31 December 2015 in one of the six university centers in the French West.

Exclusion Criteria:

* Minor patients,
* patients with a pathologic analysis in favor of a mixed secretion adenoma (positive immunohistochemical analysis for ACTH and another hormone of the anterior pituitary).
* patients who have undergone a pathologic diagnosis of "adenoma to ACTH" without clinical-biological Cushing syndrome, ie silent adenoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 at inclusion, formerly or currently being followed for Cushing's disease diagnosed between 1 January 1990 and 31 December 2015 in one of the six university centers in the French West.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Rates de remission and recurrence after the first surgery | between 1 January 1990 and 31 December 2015
  rate of postoperative 3-month remission and rate of recurrence after the first surgery

SECONDARY OUTCOMES:
predictive factors of remission and recurrence | between 1 January 1990 and 31 December 2015
  To study the significance link between the peri-operative clinical and biological characteristics and remission on the one hand and the risk of recurrence after first pituitary surgery on the other hand.